CLINICAL TRIAL: NCT05614323
Title: Eating Experience at the Comprehensive Cancer Center Wards - a Qualitative Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 202200345
Record Dates: First submitted 2022-09-12; First posted 2022-11-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Smell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Interview and determining taste and smell with taste strips and Sniffin' Sticks — The Patient-Generated Subjective Global Assessment (PG-SGA) Short Form will be filled in by the participants. Next, a semi-structured in-depth interview will be performed in a quiet environment. The interview will take a maximum of one hour and will take place once. Topics that will be discussed are eating-related problems, the taste and smell of the offered hospital food, the choice in hospital food, the ambience during the eating moments, the use of protein-enriched snacks, the difference between eating at home and at the hospital, personal tips- and-tricks to maintain adequate nutritional intake, and how patients' think that food enjoyment can be improved in the hospital. The interview will be recorded. At last, taste and smell will be objectively determined with respectively taste strips and Sniffin' Sticks.

SUMMARY:
In hospitalized patients with cancer treated with systemic therapy, semi-structured in-depth interviews will be performed. Topics that will be discussed are eating-related complaints, the taste and smell of the offered hospital food, the choice in hospital food, the ambience during the eating moments, the use of protein-enriched snacks, the difference between eating at home and at the hospital, and personal tips-and-tricks to maintain adequate nutritional intake and improve food enjoyment in the hospital. Patients will be included until data saturation is reached. The interviews will be recorded and analyzed according to the principles of thematic analysis.

DETAILED DESCRIPTION:
This qualitative study will be performed in all patients with cancer admitted to the Comprehensive Cancer Center (CCC) wards in the UMCG: medical oncology (D2) and hematology (E2). Potential participants are identified by the medical oncologists and dietitians who are part of the study team. Patients with pathologically confirmed diagnosis of all-types of cancer, treated with systemic therapy will be included. These patients are contacted during their hospital stay by their treating physician or nurse. They will introduce the study to the patient and will ask the patient permission for a visit by the investigators. The investigators will, when permission has been given, visit the patient and inform the patient about the study. Patients have to be hospitalized more than two days, as they will then have had multiple meals in a hospital environment.

Potential participants are given verbal information about the study and, if they are interested, also written study information. The potential participants are contacted by the investigators three days later for written informed consent, and setting a date for the interview, possibly during hospitalization.

At the agreed date, first, the Patient-Generated Subjective Global Assessment (PG-SGA) Short Form will be filled in by the participants. This questionnaire consists of four questions regarding weight, food intake, symptoms and activities/function. Next, a semi-structured in-depth interview will be performed in a quiet environment. The interview will take a maximum of one hour and will take place once. Topics that will be discussed are eating-related problems, the taste and smell of the offered hospital food, the choice in hospital food, the ambience during the eating moments, the use of protein-enriched snacks, the difference between eating at home and at the hospital, personal tips-and-tricks to maintain adequate nutritional intake, and how patients' think that food enjoyment can be improved in the hospital. The interview will be recorded. At last, taste and smell will be objectively determined with respectively taste strips and Sniffin' Sticks. Taste strips with an impregnated taste solution will be placed in the participants' mouth. The taste solutions contain the basic tastes bitter, sweet, sour and salty in four different concentrations, thus 16 tests will be performed. The strips will randomly be administered and participants are asked which taste they notice. A right answer gives one point and a total of 16 point can be obtained. Sniffin' Sticks are pens filled with liquid odorants, which are presented to the participants' nose. Participants will smell 16 different scents with an interval of minimal 30 seconds to prevent desensitization. For each scent, participants will choose between four options from a multiple choice card.

At last, the participants will be asked if topics were missed and if questions or topics were clear and are asked if they can be contacted for future studies. After the conversation, the background of the participant will be collected from the patients electronic file, including stage and location of primary tumor, type and status of treatment, duration of treatment, age, gender, days of hospitalization, current diet (including tube feeding and drink feeding), weight (loss), and medical history affecting taste, smell or mouthfeel.

Participants will be included until data saturation is reached, i.e., no new insights or themes are reported by the participants (15-20 participants). By purposive sampling, a varied group of participants will be included. Patients are excluded if contra-indication for oral food intake exist or oral food intake is perceived as painful by the patient. The interviews will be audio recorded, transcribed verbatim, and analyzed according to the principles of thematic analysis, with Atlas-ti. The audio recordings will be saved on the Research Drive of the UMCG and will be destroyed after transcribing. The baseline characteristics will be saved in REDCap (Research Electronic Data Capture, Version 10.0.23), an application to support data capture in a safe web-based environment, hosted by the UMCG.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of cancer
* Able to understand spoken and written Dutch
* > 18 years
* Systemic treated for cancer in a clinical setting

Exclusion Criteria:

* Contra-indication for oral food intake
* Oral food intake perceived as painful by patient
* Uncertainty about the willingness or ability of the patient to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer admitted to the Comprehensive Cancer Center wards in the UMCG: Medical Oncology and Hematology
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-11-26 (Actual)

PRIMARY OUTCOMES:
Eating experience | 11/2022 - 03/2023
  One hour interview, taste and smell tests, and answering PG-SGA questionnaire to assess eating experience (food and drinks, ambience during meals, timing of the meals, and the choice of freedom of meals) of patients with cancer admitted to the UMCG.

SECONDARY OUTCOMES:
Improving eating experience | 11/2022 - 03/2023
  One hour interview to assess possible improvements of eating experience of patients with cancer admitted to the UMCG.

CONTACTS AND LOCATIONS:
Overall Officials: Jacco J de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided